CLINICAL TRIAL: NCT05131256
Title: Neurofunctional Characterization of Emotional Regulation and Its Links With the Eating Behaviour of Patients Suffering From Obesity, With or Without Binge Eating Disorder and Seeking Bariatric Surgery. Pilot Study
Brief Title: fMRI Study of Emotion Regulation in Patients Suffering From Obesity With or Without Binge Eating Disorder and Seeking Bariatric Surgery
Acronym: OBéMO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PJ20148
Record Dates: First submitted 2021-08-03; First posted 2021-11-23 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Obesity; Binge-Eating Disorder
Keywords: Obesity; Emotion; fMRI; Emotion regulation; Binge eating disorder
MeSH Terms: conditions — Obesity; Binge-Eating Disorder; Emotional Regulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- patients suffering from obesity with BED (Experimental)
  Interventions: Behavioral: Neurofunctional characterization of emotional regulation (fMRI)
- patients suffering from obesity without BED (Active Comparator)
  Interventions: Behavioral: Neurofunctional characterization of emotional regulation (fMRI)
- healthy participants (Active Comparator)
  Interventions: Behavioral: Neurofunctional characterization of emotional regulation (fMRI)

INTERVENTIONS:
Behavioral: Neurofunctional characterization of emotional regulation (fMRI) — Investigation of neurofunctional characterization of emotional regulation and its links with the eating behaviours of patients suffering from obesity using a comprehensive, clinical, and cognitive assessment and task-based MRI exams.

SUMMARY:
Obesity is a major public health problem and Binge eating disorder (BED) is very frequently observed in patients considered for weight loss surgery and seems to influence their outcome critically. Literature highlights a global emotional overload in individuals with BED, but few are known on the mechanisms involved. The purpose of this study is to fill this gap by comparing the neurofunctional profiles of emotion regulation between patients suffering from obesity, with or without BED and healthy participants during the performance of emotion regulation tasks. Results may help to understand the neural bases of the impairments observed in patients with obesity, with or without BED, which may in turn help to propose, in the long term, potential new therapeutic approaches.

DETAILED DESCRIPTION:
Obesity is a major public health problem and frequently associated with Binge eating disorder (BED) in patients considered for weight loss surgery and seems to influence their outcome critically. It may be due, in part, to an ineffective or a maladaptive emotional regulation. Emotion regulation is the ability to exert control over one's own emotional state. The relative absence of this ability would indicate the presence of difficulties in emotion regulation, or an emotion dysregulation. Individuals with disordered eating may have a greater vulnerability to use maladaptive emotion regulation strategies. In the eating behaviours, an emotion dysregulation can cause weight gain that can lead to overweight or obesity. Accordingly, patients suffering from obesity, and with BED may have a greater vulnerability to use maladaptive emotion regulation strategies. However, few studies have investigated the neurofunctional profiles of emotion regulation in patients suffering from obesity with and without BED and seeking bariatric surgery.

The aim of the study is to explore the neural correlates of emotion regulation in patients suffering from obesity, with or without BED, in comparison with those of healthy participants. We also aim to describe the relationship between the neural correlates, eating behaviours and assessed psychological profiles.

ELIGIBILITY:
Group 1: Patients suffering from obesity, seeking bariatric surgery, and with BED.

Inclusion criteria:

* Patients between 18 and 60 years old, men or women, right-handed
* Having a diagnosis of obesity class 2 or 3 and seeking bariatric surgery
* With Binge eating disorder (BED)
* Possibility to the use of MRI
* Patients being a native French speaker
* Patients enrolled in the national healthcare insurance program
* Patients consenting to participate to the study

Exclusion criteria:

* The presence of a current substance use disorder as defined by DSM-5 criteria
* The presence of neurological disorders or head trauma
* The presence of any intellectual disability, of pervasive developmental disorders or learning difficulties (especially of dysphasia and dyspraxia)
* A current mood episode as defined by DSM-5 criteria
* A diagnosis of schizophrenia or of bipolar disorder according to DSM-5 criteria
* Handling of psychotropics substances
* A sensorial impairment uncorrected (visual and/or hearing)
* Contraindication to the use of MRI
* Pregnant woman and people particularly protected by the law

Group 2: Patients suffering from obesity, seeking bariatric surgery, and without BED.

Inclusion criteria:

* Patients between 18 and 60 years old, men or women, right-handed
* Having a diagnosis of obesity class 2 or 3 and seeking bariatric surgery
* Without Binge eating disorder (BED)
* Possibility to the use of MRI
* Patients being a native French speaker
* Patients enrolled in the national healthcare insurance program
* Patients consenting to participate to the study

Exclusion criteria:

* The presence of a current substance use disorder as defined by DSM-5 criteria
* The presence of neurological disorders or head trauma
* The presence of any intellectual disability, of pervasive developmental disorders or learning difficulties (especially of dysphasia and dyspraxia)
* A current mood episode as defined by DSM-5 criteria
* A diagnosis of schizophrenia or of bipolar disorder according to DSM-5 criteria
* Handling of psychotropics substances
* A sensorial impairment uncorrected (visual and/or hearing)
* Contraindication to the use of MRI
* Pregnant woman and people particularly protected by the law

Group 3: Healthy participants.

Inclusion criteria:

* Men or women, right-handed, between 18 and 60 years old
* Without overweight nor obesity
* Native French speaker
* Individuals enrolled in the national healthcare insurance program
* Individuals consenting to participate to the study

Exclusion criteria:

* Past obesity
* The presence of neurological disorders or head trauma
* The presence of any intellectual disability, of pervasive developmental disorders or learning difficulties (especially of dysphasia and dyspraxia)
* Handling of psychotropics substances
* A sensorial impairment uncorrected (visual and/or hearing)
* Contraindication to the use of MRI
* Pregnant woman and people particularly protected by the law
* A current mood episode as defined by DSM-5 criteria
* A diagnosis of schizophrenia or of bipolar disorder according to DSM-5 criteria
* The presence of a current substance use disorder as defined by DSM-5 criteria
* A diagnosis of eating disorder as defined by DSM-5 criteria

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-07-20 (Actual); Primary Completion 2025-07-20 (Estimated); Study Completion 2025-07-20 (Estimated)

PRIMARY OUTCOMES:
fMRI activations during an emotional regulation task (a cognitive reappraisal task) | Day 0
  The participant either reappraises or passively watches negative or neutral pictures and rates his affect (visual analogue scale: 0 to 10, high scores mean negative feelings).
fMRI activations during the inhibition of an ongoing motor response under an emotional condition (emotional stop signal task) | Day 0
  The participant is presented with a series of images comprised of neutral, positive, and negative categories and is instructed to categorize the images according to their valence (Go trials). Some trials include a stop signal indicating that the participant should inhibit his behavioral response and associated emotional reaction (Stop trials).
fMRI activations during the performance of an emotion regulation task (an emotional Stroop task) | Day 0
  The participant is asked to count how many numbers are presented on the screen. Numbers may match the value of the number (congruent condition) or not (incongruent condition). The numbers are preceded by emotional stimuli (negative, positive, neutral). The participant also views the emotional stimuli pictures without counting numbers (view condition).

SECONDARY OUTCOMES:
Description of eating behaviours: Binge eating | Day 0
  The Binge Eating Scale (BES) is a 16-item self-administered questionnaire used to assess the presence of binge eating behavior indicative of an eating disorder. Eight items describe behavioral manifestations (for example, eating fast or consuming large amounts of food) and eight items on associated feelings and cognitions (for example, fear of not stopping eating). Each item has a response range from 0 to 3 points (0 = no severity of the BES symptoms, 3 = serious problems on the BES symptoms). Marcus et al. (1988) created a range of scores for the BES from 0 to 46 points: a score of less than 17 points indicates minimal binge eating (BE) problems; a score between 18 and 26 points indicates moderate BE problems, and a score of more than 27 points indicates severe BE problems. We consider binge eating as a categorical variable (significant binge eating if BES score ≥18).
Description of eating behaviours: Emotional eating, external eating, restraint eating | Day 0
  The Dutch Eating Behavior Questionnaire (DEBQ) is administered using the French version to assess three components of eating behavior: emotional, external, and restrained eating. It is a self-report measure that contains 33 items. Thirteen items assess emotional eating, 10 items assess external eating, and 10 items assess restrained eating. Each item is rated on a 5-point Likert scale. Higher scores on each dimension mean worse eating behaviors.
Description of eating behaviours: Bulimic symptomatology | Day 0
  The Bulimic Investigatory Test, Edinburgh (BITE) is a self-report questionnaire used to evaluate the presence and severity of bulimic symptomatology. It is composed of 33 items divided into two different subscales: a symptom subscale (30 items) and a severity subscale (3 items). Henderson and Freeman (1987) considered a BITE score under 10 points as indicative of no problem with eating behavior, a score between 10 and 20 points as indicative of abnormal eating patterns (from 15 to 20 points warns us of the presence of a possible subthreshold bulimia nervosa), and a score higher than 20 points constitutes altered eating patterns with a possible bulimia nervosa.
Description of psychological profiles (emotional, cognitive and personality): Emotion regulation | Day 0
  The Difficulty in Emotion Regulation Scale (DERS) is a 36-item self-report questionnaire. It assesses six different aspects of emotional regulation including non-acceptance of emotional responses (Non-Acceptance), difficulty engaging in goal-directed behavior (Goals), impulse control difficulties (Impulse), lack of emotional awareness (Awareness), limited access to emotional regulation strategies (Strategies), and lack of emotional clarity (Clarity). Higher scores on each dimension indicate greater emotion dysregulation symptoms.
Description of psychological profiles (emotional, cognitive and personality): Depression severity | Day 0
  Depression severity is assessed with the shortened Beck Depression Inventory (BDI). This is a widely used self-report scale consisting of 13 items, which has been validated in French. The total score is obtained by adding the scores of the 13 items and ranges from 0 to 39, with higher scores indicating greater depression symptoms.
Description of psychological profiles (emotional, cognitive and personality): Anxiety severity | Day 0
  Anxiety severity is assessed with the Spielberger State-Trait Inventory (STAI) which is a 40-item scale, using a 4-point Likert scale for each item. This scale was used to measure both trait anxiety (how dispositionally anxious a person is across time and situations) and state anxiety (how anxious a person is feeling at a particular moment). Higher scores indicate greater anxiety symptoms.
Description of psychological profiles (emotional, cognitive and personality): Impulsivity | Day 0
  We use the UPPS-P Impulsive Behavior Scale to assess the facets of impulsivity, i.e., Negative Urgency, Positive Urgency, (lack of) Premeditation, (lack of) Perseverance, and Sensation Seeking. This shortened version (20 items) has 4 items per scale, and each item is responded to on a 4-point Likert-type scale. Higher scores on each scale indicate greater impulsivity symptoms. This self-report scale has received endorsement from the National Institutes of Health's (NIH) PhenX Toolkit as the recommended self-report measure of impulsigenic traits.

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France